CLINICAL TRIAL: NCT03186209
Title: A Multicentre, Randomised, Double-blind, Parallel Group, Placebocontrolled, Phase 3 Efficacy and Safety Study of Benralizumab (MEDI-563) Added to Medium to High-dose Inhaled Corticosteroid Plus Long-acting β2 Agonist in Patients With Uncontrolled Asthma.
Brief Title: Efficacy and Safety Study of Benralizumab in Patients With Uncontrolled Asthma on Medium to High Dose Inhaled Corticosteroid Plus LABA (MIRACLE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D3250C00036; 2017-000702-38 (EudraCT Number)
Record Dates: First submitted 2017-05-19; First posted 2017-06-14 (Actual); Results first posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-03

CONDITIONS: Asthma
Keywords: Asthma,; Bronchial Diseases,; Respiratory Tract Diseases,; Lung Diseases,; Obstructive Lung Diseases
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Benralizumab (Experimental): Benralizumab administered subcutaneously
  Interventions: Biological: Benralizumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab subcutaneously on study week 0 until study week 40 inclusive.
  Arms: Benralizumab
Biological: Placebo — Placebo subcutaneously on study week 0 until study week 40 inclusive.
  Arms: Placebo

SUMMARY:
This is a randomised, double-blind, parallel group, placebo-controlled study designed to evaluate the efficacy and safety of a fixed 30 mg dose of benralizumab administered subcutaneously for patients with a history of asthma exacerbations and uncontrolled asthma receiving medium to high-dose inhaled corticosteroid plus long-acting β2-agonist (ICS-LABA) with or without oral corticosteroids and additional asthma controllers.

DETAILED DESCRIPTION:
Approximately 666 patients will be randomised. Patients will be stratified by country/region, age group (adult or adolescent), and peripheral blood eosinophil count at time of Visit 1 (<300 or ≥300 cells/μL).All the patients will be randomised to either placebo or benralizumab (1:1 ratio) for a 48-weeks treatment, every 4 weeks for the first 3 doses and then every 8 weeks thereafter.

ELIGIBILITY:
Key Inclusion Criteria:

1. Written informed consent, and assent when applicable for study participation must be obtained prior to any study related procedures being performed (local regulations are to be followed in determining the assent/consent requirements for children and parent[s]/guardian[s]) and according to international guidelines and/or applicable local guidelines.
2. Female and male aged 12 to 75 years, inclusively, at the time of Visit 1. For those patients, who are 17 on the day of Visit 1 but will turn 18 after this day, will be considered an adolescent for the purposes of this trial.
3. History of physician-diagnosed asthma requiring treatment with medium-to-high dose ICS (>250μg fluticasone propionate dry powder formulation equivalents total daily dose) and a LABA, for at least 6 months prior to Visit 1.
4. Additional maintenance asthma controller medications that are locally approved in a country for the treatment of asthma (e.g., leukotriene receptor antagonists (LTRAs), tiotropium, chromone, theophylline, oral corticosteroid), and have been used for at least 30 days prior to Visit 1 are allowed.
5. At least 2 documented asthma exacerbations in the 12 months prior to the date informed consent, and assent when available, during the treatment of medium-to-high dose ICS-LABA that required use of a systemic corticosteroid or a temporary increase from the patient's usual maintenance dose of oral corticosteroid. For patients who are re-screened within 30 days of their screen failure date, the calculation of the 12 month period should be done from the original informed consent, and assent when applicable date.
6. Documented post-bronchodilator (post-BD) reversibility in FEV1 of >12% and >200 mL in FEV1 within 12 months prior to Visit 1. If historical documentation is not available, reversibility must be demonstrated and documented at Visit 2.
7. Fulfilment of at least 1 of the following conditions over the 7 days prior to randomization:

   * >2 days with a daytime or night time symptoms score >1
   * Rescue Short-acting β2 agonist (SABA) use on >2 days
   * ≥1 nocturnal awakening due to asthma
8. Pre-bronchodilator (Pre-BD) FEV1 of <80% predicted (<90% predicted for patients aged 12 to 17 years) at Visit 2.
9. ACQ-6 score > = 1.5 at Visit 2.

Exclusion Criteria:

1. Known history of clinically important pulmonary disease other than asthma (e.g., active lung infection, chronic obstructive pulmonary disease (COPD), bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (e.g,. allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
2. Known history of any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, haematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the studies or their interpretations
   * Impede the patient's ability to complete the entire duration of study.
3. Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent, and assent when applicable, is obtained or during the screening period.
4. Any clinically significant abnormal findings in physical examination, vital signs, haematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study.
5. Current smokers or former smokers with a smoking history of > 10 pack-years.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 695 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- China (34):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Changzhi
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Foshan
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hohhot
  - Research Site, Jining
  - Research Site, Kunming
  - Research Site, Lishui
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Neijiang
  - Research Site, Qingdao
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Taiyuan
  - Research Site, Taizhou
  - Research Site, Wanzhou
  - Research Site, Wuhan
  - Research Site, Xiangtan
  - Research Site, Xinxiang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
  - Research Site, Zhuhai
  - Research Site, Zunyi
- Philippines (2):
  - Research Site, Iloilo City
  - Research Site, Manila
- South Korea (10):
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheonan
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
- Taiwan (2):
  - Research Site, Taipei
  - Research Site, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Jin Y, Guiastrennec B, Stuke M, Yao Y, Zhang Y, Barker P, Jison M, Penland RC, Ding J, Lukka PB. Population Pharmacokinetics and Exposure-Response Analysis of Benralizumab in Chinese Adults, Adolescents, and Pediatric Participants with Severe Eosinophilic Asthma. Clin Pharmacokinet. 2025 Aug;64(8):1231-1243. doi: 10.1007/s40262-025-01538-9. Epub 2025 Jun 23. PMID 40551003
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00036&attachmentIdentifier=94f140e1-8d12-441f-a36f-47b7a861e52c&fileName=5Sep2023-d3250c00036-csp-v5_Redacted_.pdf&versionIdentifier=
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00036&attachmentIdentifier=cc47324b-7f06-401d-a8ed-a6a71fd95944&fileName=d3250c00036-sap-ed3_Redacted_5Sep2023.pdf&versionIdentifier=
- See also: Redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D3250C00036&attachmentIdentifier=2640ddf4-529a-41b1-877d-3d53a0495d8a&fileName=d3250c00036-study-synopsis_Redacted_5Sep2023.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 695 participants were randomized to receive treatment in study D3250C00036 (MIRACLE) with Benralizumab or placebo. All the 695 randomized participants received treatment with study drug.
Pre-assignment Details: At the first visit, ie, the enrollment visit 1, participants were evaluated regarding the protocol mandated inclusion and exclusion criteria. After enrollment, eligible participants were randomized to either placebo or Benralizumab 30 mg at a 1:1 ratio, administered subcutaneously every 4 weeks for the first 3 doses and then every 8 weeks thereafter.
Groups:
- Benralizumab 30 mg: Benralizumab administered subcutaneously
Period: Overall Study
Arm/Group | Benralizumab 30 mg | Placebo
Started (All Participants Randomized) | 348 | 347
Dosed (Full Analysis Set) | 348 | 347
Completed (study) | 331 | 321
Not Completed | 17 | 26
Not completed — Withdrawal by Subject | 11 | 22
Not completed — Pregnancy | 1 | 0
Not completed — Adverse Event | 4 | 0
Not completed — V18 SKIPPED DUE TO LOGISTICS REASON | 1 | 0
Not completed — PI DECIDED TO DISCONTINUE THE STUDY DUE TO THE LACK OF CRC RESOURCES | 0 | 2
Not completed — Fail to meet randomization criteria | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set, all participants who were randomized and received at least one investigational product (IP), Benralizumab or Placebo.
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg | Placebo | Total
Number analyzed (Participants) | 348 | 347 | 695
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (11.56) | 51.0 (12.56) | 51.1 (12.06)
Age, Customized [Number; unit: Participants]
  >=12 - <18 years | 1 | 0 | 1
  >=18 - <65 years | 299 | 295 | 594
  >=65 - <=75 | 48 | 52 | 100
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 221 | 207 | 428
  Male | 127 | 140 | 267
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Non-Hispanic or Latino | 348 | 347 | 695
  Asian | 348 | 347 | 695

OUTCOME MEASURES:

1. Primary Outcome: Annual Asthma Exacerbation Rate in Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma for Baseline Eosinophils >=300/uL
Description: Annual asthma exacerbation rate over the 48-week treatment period among benralizumab and placebo groups
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: events/patient-year
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 236 | 237
events/patient-year | 0.49 [0.33 to 0.72] | 1.88 [1.35 to 2.61]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Negative binomial — Multiplicity protected by hierarchy testing procedure. First in line hypothesis testing, requiring p-value <0.05; Model with covariates: treatment group, region (China/Non-China), number of exacerbations in previous year, use of maintenance oral corticosteroids; Rate Ratio = 0.26, 95% CI 2-sided [0.19 to 0.36]

2. Secondary Outcome: Change From Baseline at Week 48 in Pre-bronchodilator FEV1 (L) Value for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Change from baseline at Week 48 in Pre-bronchodilator FEV1 (L)
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL; number analyzed refers to records with value available at Week 48 for this outcome measure
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 215 | 204
Liter | 0.333 (0.4499) | 0.103 (0.4841)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Test after significant primary endpoint. Two secondary endpoints (change in FEV1 and total asthma symptom score) using Holm's procedure; smaller p-value to be <0.025, and larger p-value to be <0.05; Model includes Treatment, baseline pre-bronchodilator FEV1, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [0.17 to 0.34]

3. Secondary Outcome: Change From Baseline at Week 48 in Total Asthma Symptom Score for for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Daytime and nighttime symptoms are reported using a response scale ranging from 0 to 3 where 0 indicates no asthma symptoms. The total asthma symptom score is the sum of the daytime and nighttime scores and ranges from 0 to 6; a decrease in score indicates symptom improvement.
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 213 | 206
Scores on a scale | -1.07 (1.126) | -0.80 (1.129)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0126, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Model includes Treatment, baseline total asthma symptom score, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.45 to -0.05]

4. Secondary Outcome: Change From Baseline at Week 48 in Total Asthma Rescue Medication Use for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Change from baseline at week 48 in total rescue medication use (number of puffs/day)
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Puffs/day
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 213 | 206
Puffs/day | -0.85 (1.865) | -0.89 (2.213)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.1835, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; Model includes Treatment, baseline total asthma rescue medication use, region, use of maintenance oral corticosteroids, visit, treatment*visit; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.42 to 0.08]

5. Secondary Outcome: Change From Baseline at Week 48 in Morning Peak Expiratory Flow (PEF) for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Change from baseline at week 48 in morning PEF
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 213 | 207
L/min | 54.194 (86.3963) | 12.995 (68.7947)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; Model includes Treatment, baseline morning PEF, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = 38.66, 95% CI 2-sided [24.24 to 53.07]

6. Secondary Outcome: Change From Baseline at Week 48 in Evening Peak Expiratory Flow (PEF) for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Change from baseline at week 48 in evening PEF
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 217 | 209
L/min | 45.661 (85.4642) | 7.989 (68.0632)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; Model includes Treatment, baseline evening PEF, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = 35.85, 95% CI 2-sided [21.52 to 50.18]

7. Secondary Outcome: Change From Baseline at Week 48 in the Proportion of Night Awakening Due to Asthma and Requiring Rescue Medication for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Change from baseline at Week 48 in proportion of night awakening due to asthma and requiring rescue medication
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 217 | 208
Proportion of nights | -0.15 (0.220) | -0.15 (0.260)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.3385, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; Model includes Treatment, baseline proportion of nights awakening, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.03 to 0.01]

8. Secondary Outcome: Change From Baseline at Week 48 in Asthma Control Questionnaire 6 (ACQ-6) for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: ACQ-6 contains one bronchodilator question and 5 symptom questions. Questions are rated from 0 (totally controlled) to 6 (severely uncontrolled). Mean ACQ-6 score is the average of the responses.
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 218 | 212
Scores on a scale | -1.22 (0.901) | -0.79 (0.962)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; Model includes Treatment, baseline ACQ-6 score, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-0.58 to -0.28]

9. Secondary Outcome: Time to First Asthma Exacerbation for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Time to first asthma exacerbation over 48-week treatment period
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 236 | 237
Days | NA [NA to NA] — The number of exacerbations is small, thus the Median survival time to first exacerbation has not reached. | 227 [146 to NA] — Insufficient number of exacerbations to estimate upper limit of 95% CI.
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Regression, Cox — Nominal p-value. Not multiplicity protected by testing procedure; model including covariates treatment group, region, number of exacerbations in the previous year, and use of maintenance oral corticosteroids; Hazard Ratio (HR) = 0.32, 95% CI 2-sided [0.23 to 0.43]

10. Secondary Outcome: Number and Percentage of Patients With >=1 Asthma Exacerbations Among Patients Who Were on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Number and percentage of patients with at least one exacerbation over 48-week treatment period
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 236 | 237
Participants | 55 | 125
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Nominal p-value. Not multiplicity protected by testing procedure; Controlling for region, number of exacerbations in the previous year (2, >=3), use of OCS; Odds Ratio (OR) = 0.28, 95% CI 2-sided [0.19 to 0.42]

11. Secondary Outcome: Change From Baseline at Week 48 in Total Score of St. George's Respiratory Questionnaire (SGRQ) for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: The SGRQ is a 50-item PRO instrument developed to measure the HRQoL of patients with airway diseases. The questionnaire is divided into two parts: part 1 consists of 8 items pertaining to the severity of respiratory symptoms in the preceding 4 weeks; part 2 consists of 42 items related to the daily activity and psychosocial impacts of the individual's respiratory condition. The total score indicates the impact of disease on overall HRQoL. This total score is expressed as a percentage of overall impairment, in which 100 represents the worst possible HRQoL and 0 indicates the best possible HRQoL.
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 209 | 200
Scores on a scale | -23.24 (20.509) | -14.75 (21.838)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; Model with covariates: treatment group, baseline SGRQ total score, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = -9.19, 95% CI 2-sided [-12.79 to -5.60]

12. Secondary Outcome: Annual Asthma Exacerbation Rate Associated With an Emergency Room/Urgent Care Visit or a Hospitalization for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Annual asthma exacerbation rate associated with an emergency room/urgent care visit or a hospitalization over 48-week treatment period
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: events/patient-year
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 236 | 237
events/patient-year | 0.06 [0.04 to 0.11] | 0.14 [0.09 to 0.20]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0222, Negative binomial — Nominal p-value. Not multiplicity protected by testing procedure; Model includes Treatment, use of maintenance oral corticosteroids, categorical variable of ER/UC or hospitalization exacerbations during previous year; Rate ratio = 0.46, 95% CI 2-sided [0.24 to 0.90]

13. Secondary Outcome: Number and Percentages of Asthma Specific Health Care Resource Utilization for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Asthma specific health care resource utilization over 48-week treatment period.
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils >=300/uL
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 236 | 237
Participants
  Hospitalisations | 6 | 21
  Emergency Department Visits | 11 | 12
  Unscheduled Outpatient Visits | 53 | 99
  Home Visits | 1 | 2
  Telephone Calls | 35 | 71
  Ambulance Transports | 2 | 2
  Advanced Pulmonary Function Test | 4 | 8

14. Secondary Outcome: The Pharmacokinetics (PK) of Benralizumab as Assessed by Trough Concentration
Description: PK trough concentrations at each visit
Time Frame: week 0, week 24, week 48
Population: PK analysis set; number analyzed includes participants with available value at each specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 345 | 0
ng/mL
  Week 0 | 0 (0) |
  Week 24: number analyzed (Participants) | 297 | 0
  Week 24 | 137.914 (432.419) |
  Week 48: number analyzed (Participants) | 289 | 0
  Week 48 | 123.476 (395.951) |

15. Secondary Outcome: The Immunogenicity of Benralizumab as Assessed by the Presence of Anti-drug Antibodies (ADAs)
Description: Anti-drug antibodies (ADA) responses at baseline and post baseline.
Time Frame: Pre-treatment until end of 48-week end of treatment
Population: Safety analysis set; number analyzed includes participants with available value at each specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 348 | 347
Participants
  ADA positive at any time, including baseline and/or post-baseline (ADA prevalence) | 58 | 6
  Treatment-emergent ADA positive, including treatment-induced and treatment-boosted ADA positive: number analyzed (Participants) | 345 | 347
  Treatment-emergent ADA positive, including treatment-induced and treatment-boosted ADA positive | 58 | 2
  Treatment-induced ADA positive: number analyzed (Participants) | 345 | 336
  Treatment-induced ADA positive | 56 | 2
  Treatment-boosted ADA positive: number analyzed (Participants) | 345 | 336
  Treatment-boosted ADA positive | 2 | 0
  ADA positive at both baseline and at least one post-baseline assessment: number analyzed (Participants) | 345 | 336
  ADA positive at both baseline and at least one post-baseline assessment | 2 | 2
  ADA positive at baseline only | 0 | 2
  ADA persistently positive: number analyzed (Participants) | 345 | 336
  ADA persistently positive | 40 | 1
  ADA transiently positive: number analyzed (Participants) | 345 | 336
  ADA transiently positive | 16 | 1
  ADA positive with maximum titre > median of maximum titres | 25 | 2
  ADA positive with maximum titre <= median of maximum titres | 33 | 4
  nAb prevalence (nAb positive at any time, including baseline and/or post-baseline) | 55 | 1
  nAb incidence: number analyzed (Participants) | 345 | 336
  nAb incidence | 55 | 1

16. Secondary Outcome: Percent Change From Baseline at Week 48 in Blood Eosinophil Levels for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils >=300/uL
Description: Percent change from baseline at Week 48 in blood eosinophil levels
Time Frame: From randomization through Study Week 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 213 | 199
Percent change | -80.6 (34.65) | 42.3 (380.86)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p < 0.0001, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; model includes treatment , baseline eosinophil count, region, use of maintenance oral corticosteroids, visit, and treatment by visit; Mean Difference (Final Values) = -119.31, 95% CI 2-sided [-169.78 to -68.84]

17. Other Pre Specified Outcome: Annual Asthma Exacerbation Rate in Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils <300/uL
Description: Annual asthma exacerbation rate over the 48-week treatment period among benralizumab and placebo groups
Time Frame: From randomization through Study Week 48.
Population: Full analysis set, Baseline eosinophils <300/uL
Measure: Least Squares Mean (95% Confidence Interval); unit: events/patient-year
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 112 | 110
events/patient-year | 0.72 [0.49 to 1.06] | 0.87 [0.61 to 1.24]
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.4519, Negative binomial — Nominal p-value. Not multiplicity protected by testing procedure; [statistical method as in outcome 1, analysis 1]; Rate Ratio = 0.83, 95% CI 2-sided [0.51 to 1.35]

18. Other Pre Specified Outcome: Change From Baseline at Week 48 in Pre-bronchodilator FEV1 (L) Value for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils <300/uL
Description: Change from baseline at Week 48 in Pre-bronchodilator FEV1 (L)
Time Frame: From randomization through Study Week 48
Population: Full analysis set, Baseline eosinophils <300/uL; number analyzed refers to records with value available at Week 48 for this outcome measure
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 101 | 97
Liter | 0.178 (0.4068) | 0.045 (0.3626)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.0214, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.12, 95% CI 2-sided [0.02 to 0.22]

19. Other Pre Specified Outcome: Change From Baseline at Week 48 in Total Asthma Symptom Score for Patients on Medium to High-dose ICS-LABA With Uncontrolled Asthma and Baseline Eosinophils <300/uL
Description: as for outcome 3
Time Frame: From randomization through Study Week 48
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg | Placebo
Number analyzed (Participants) | 101 | 94
Scores on a scale | -0.97 (1.260) | -0.75 (1.105)
Statistical Analysis 1: Comparison: Benralizumab 30 mg vs Placebo; Test type: Superiority; p = 0.1589, Mixed Models Analysis — Nominal p-value. Not multiplicity protected by testing procedure; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.51 to 0.08]

ADVERSE EVENTS:
Time Frame: From initial dose of the study treatment to the end of study, i.e., up to 56 weeks of follow-up.
Description: All treated participants from the first dose to the end of study. Total of 695 participants with 348 participants treated with Benralizumab administered every 4 weeks for the first 3 doses and then every 8 weeks and 347 were under placebo treatment.
Arm/Group | Benralizumab 30 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/348 | 0/347
Serious Adverse Events (participants affected / at risk) | 44/348 | 63/347
Other Adverse Events (participants affected / at risk) | 194/348 | 194/347
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg (N=348) | Placebo (N=347)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0)
Reflux gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 1 (1) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis allergic (Infections and infestations) | 1 (1) | 0 (0)
Chronic sinusitis (Infections and infestations) | 2 (2) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4) | 6 (6)
Pneumonia bacterial (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenolymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 33 (37)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Neurogenic shock (Vascular disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg (N=348) | Placebo (N=347)
Pyrexia (General disorders) | 18 (22) | 9 (9)
Bronchitis (Infections and infestations) | 11 (15) | 27 (40)
COVID-19 (Infections and infestations) | 11 (11) | 6 (6)
Nasopharyngitis (Infections and infestations) | 28 (36) | 33 (48)
Otitis media (Infections and infestations) | 11 (11) | 8 (9)
Pharyngitis (Infections and infestations) | 13 (13) | 13 (14)
Pneumonia (Infections and infestations) | 9 (13) | 16 (19)
Rhinitis (Infections and infestations) | 13 (14) | 6 (9)
Upper respiratory tract infection (Infections and infestations) | 120 (200) | 120 (230)
Urinary tract infection (Infections and infestations) | 9 (10) | 12 (14)
Dizziness (Nervous system disorders) | 11 (11) | 8 (14)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 22 (41) | 15 (17)
Hypertension (Vascular disorders) | 7 (7) | 13 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and/or the Principal Investigator shall not include in or shall remove from any proposed publication any Confidential Information, errors or inaccuracies; and shall withhold publication, submission for publication or presentation for a period of ninety (90) days from the date on which the Company receives the material to allow the Company to take such measures as the Company considers necessary to preserve its proprietary rights and/or protect its Confidential Information.

DOCUMENTS (2):
  • Study Protocol (2020-12-18): https://cdn.clinicaltrials.gov/large-docs/09/NCT03186209/Prot_000.pdf
  • Statistical Analysis Plan (2023-01-31): https://cdn.clinicaltrials.gov/large-docs/09/NCT03186209/SAP_001.pdf